CLINICAL TRIAL: NCT05835765
Title: Use of Dynamic Elastometric Body in Preterm Newborns: A Prospective Pilot Study With a Medical Device
Brief Title: Use of Dynamic Elastometric Body in Preterm Newborns
Acronym: BODYNEO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Romeo Domenico Marco, Assistant professor, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5364
Record Dates: First submitted 2023-03-28; First posted 2023-04-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Premature Birth
Keywords: prematurity; Hyperexcitability syndrome; Neonatal intensive care; Dynamic Elastometric device
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic Elastometric Body and neurological evaluation (Experimental): Use of dynamic elastometric body for one week and neurological evaluation before use of body, at 30 minutes after application, at one week after using the device and at 1th months since discharge
  Interventions: Device: Dynamic Elastometric Body in Preterm Newborns
- Neurological evaluation (No Intervention): Neurological evaluation at enrollment, at one week after enrollment and at 1th months since discharge

INTERVENTIONS:
Device: Dynamic Elastometric Body in Preterm Newborns — The study group made up of 12 newborns will use Flexa bodysuits made to the measurements of newborns.The bodysuit will be worn for a minimum of 4 hours and a maximum of 6 hours each day for a week (depending on any signs of discomfort). After 6 hours, the body will be removed and reapplied the next day for 4-6 hours. The child will use the same leotard for the entire study period (1 week) and changed only if dirty.
  Arms: Dynamic Elastometric Body and neurological evaluation

SUMMARY:
The goal of this prospective pilot study is to test the use of dynamic elastomeric body in a population of preterm newborns with hyperexcitability syndrome.

The main questions it aims to answer are:

* To evaluate the effectiveness of the body in elasto-compressive material (FLEXA) in addition to standard care;
* To evaluate how the use of dynamic elastomeric body promote postural containment, reduce hyperexcitability (tremor and crying), improve the organization of movement and reduce respiratory distress.

Participants will be given to routine clinical evaluations that are part of the standard of care of the premature infant admitted to Neonatology.

The clinical evaluation shall consist of:

* Hammersmith neonatal neurological examination;
* Neonatal Intensive Care Unit Network Neurobehavioural Scale (NNNS);
* General Movement's (GM's)
* Goal Attainment Scaling (GAS) Researchers will compare a study group that will be subjected to treatment with the body in elasto-compressive material and a control group without using the body in elasto-compressive material.

ELIGIBILITY:
Inclusion Criteria:

* Signs of hyperexcitability such as tremors, sudden and chaotic movements, prevalent extensor tone, postural instability and/or neurovegetative phenomena;
* Low neurological risk, i.e., according to the protocols implemented in the standard clinical practice of the Neonatology unit, a cerebral ultrasound is performed for those born between 28-32 weeks of GA, and for those born before 28 weeks of GA, an MRI of the brain) from which it may derive;
* Cerebral ultrasound normal or with minor ultrasound findings such as grade 1 intraventricular hemorrhage (germinal matrix hemorrhage with intraventricular hemorrhage covering less than 10% of the ventricular area in the parasagittal window), or evidence of transient focal white matter hyperechogenicity.
* Issue of informed consent by the parent or legal guardian.

Exclusion Criteria:

* Neuroimaging findings of major brain lesions, such as evidence of grade 2 or greater intraventricular hemorrhage on cerebral ultrasonography (germinal matrix hemorrhage with intraventricular hemorrhage over 10% of the ventricular area in the parasagittal window/with periventricular hyperechogenicity ) or persistent hyperechogenicity for more than a week;
* Presence of: ongoing infectious states and/or sepsis, ostomy wearers, severe cardio-respiratory disorders at the time of enrolment; diagnosis of genetic or metabolic diseases; carriers of cerebral malformations; invasive or non-invasive respiratory assistance;
* Failure to issue informed consent by the parent or legal guardian.

Ages: 8 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Modification or reduction of hyperexcitability syndrome with the use of Dynamic Elastometric Bodysuit | baseline
  Modification or reduction of hyperexcitability syndrome with use of Dynamic Elastometric Bodysuit in addition to standard care in terms of improvement of Goal Attainment Scaling (GAS) between the two groups. The GAS scale report a 5 level score between -2 ( worse score) to +2 (better score)
Modification or reduction of hyperexcitability syndrome with the use of Dynamic Elastometric Bodysuit | One week of application of Dynamic Elastometric Body
  Modification or reduction of hyperexcitability syndrome with use of Dynamic Elastometric Bodysuit in addition to standard care in terms of improvement of Goal Attainment Scaling (GAS) between the two groups. The GAS scale report a 5 level score between -2 ( worse score) to +2 (better score)
Modification or reduction of hyperexcitability syndrome with the use of Dynamic Elastometric Bodysuit | at one month from hospital discharge
  Modification or reduction of hyperexcitability syndrome with use of Dynamic Elastometric Bodysuit in addition to standard care in terms of improvement of Goal Attainment Scaling (GAS) between the two groups. The GAS scale report a 5 level score between -2 ( worse score) to +2 (better score)

SECONDARY OUTCOMES:
Neurological Outcome with Hammersmith neonatal neurological examination (HNNE) | baseline
  Differences in neurological evaluation indices carried out with Hammersmith neonatal neurological examination between the two groups. The HNNE report a score between 0 and 34; scores >30.5 are considered normal.
Neurological Outcome with Hammersmith neonatal neurological examination (HNNE) | One week after the use of Dynamic Elastometric Body
  Differences in neurological evaluation indices carried out with Hammersmith neonatal neurological examination between the two groups. The HNNE report a score between 0 and 34; scores >30.5 are considered normal.
Neurological Outcome with Hammersmith neonatal neurological examination (HNNE) | At one month from hospital discharge
  Differences in neurological evaluation indices carried out with Hammersmith neonatal neurological examination between the two groups. The HNNE report a score between 0 and 34; scores >30.5 are considered normal.
Neurobehavioural Outcome with NICU Network Neurobehavioural Scale (NNNS). | baseline
  Differences in neurological evaluation indices carried out with NICU Network Neurobehavioural Scale between the two group. The NNNS considering the 10th and 90th percentiles as cutoff points for normative performance.
Neurobehavioural Outcome with NICU Network Neurobehavioural Scale (NNNS). | One week after the use of Dynamic Elastometric Body
  Differences in neurological evaluation indices carried out with NICU Network Neurobehavioural Scale between the two groups. The NNNS considering the 10th and 90th percentiles as cutoff points for normative performance.
Neurobehavioural Outcome with NICU Network Neurobehavioural Scale (NNNS). | At one month from hospital discharge
  Differences in neurological evaluation indices carried out with NICU Network Neurobehavioural Scale between the two groups. The NNNS considering the 10th and 90th percentiles as cutoff points for normative performance.
Neurological Outcome with "Prechtl's Assessment of General Movements (GMs)" | baseline
  Differences in neurological evaluation indices carried out with General movements between the two groups. The GMs report a classification in: normal writhing, poor repertoire, cramped synchronised and chaotic. The classification considering cramped synchronised and chaotic movements pathological.
Neurological Outcome with "Prechtl's Assessment of General Movements (GMs)" | One week after the use of Dynamic Elastometric Body
  Differences in neurological evaluation indices carried out with General movements between the two groups. The GMs report a classification in: normal writhing, poor repertoire, cramped synchronised and chaotic. The classification considering cramped synchronised and chaotic movements pathological.
Neurological Outcome with "Prechtl's Assessment of General Movements (GMs)" | At one month from hospital discharge
  Differences in neurological evaluation indices carried out with General movements between the two groups. The GMs report a classification in: normal writhing, poor repertoire, cramped synchronised and chaotic. The classification considering cramped synchronised and chaotic movements pathological.
Neurological Outcome with "Prechtl's Assessment of General Movements (GMs)" | At 30 minutes from the use of Dynamic Elastometric Body
  Evaluation of the variation of neurological evaluation indices carried out with General movements in the study group. The GMs report a classification in: normal writhing, poor repertoire, cramped synchronised and chaotic. The classification considering cramped synchronised and chaotic movements pathological.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli -IRRCS, Rome, Italy

REFERENCES:
- [Background] Tognetti A, Lorussi F, Tesconi M, Bartalesi R, Zupone G, De Rossi D. Wearable kinesthetic systems for capturing and classifying body posture and gesture. Conf Proc IEEE Eng Med Biol Soc. 2005;2006:1012-5. doi: 10.1109/IEMBS.2005.1616589. PMID 17282358
- [Background] Matthews MJ, Watson M, Richardson B. Effects of dynamic elastomeric fabric orthoses on children with cerebral palsy. Prosthet Orthot Int. 2009 Dec;33(4):339-47. doi: 10.3109/03093640903150287. PMID 19961295
- [Background] Watson MJ, Crosby P, Matthews M. An evaluation of the effects of a dynamic lycra orthosis on arm function in a late stage patient with acquired brain injury. Brain Inj. 2007 Jun;21(7):753-61. doi: 10.1080/02699050701481613. PMID 17653949
- [Background] Cholewicki J, Lee AS, Peter Reeves N, Morrisette DC. Comparison of trunk stiffness provided by different design characteristics of lumbosacral orthoses. Clin Biomech (Bristol). 2010 Feb;25(2):110-4. doi: 10.1016/j.clinbiomech.2009.10.010. Epub 2009 Dec 9. PMID 20004503
- [Background] Flanagan A, Krzak J, Peer M, Johnson P, Urban M. Evaluation of short-term intensive orthotic garment use in children who have cerebral palsy. Pediatr Phys Ther. 2009 Summer;21(2):201-4. doi: 10.1097/PEP.0b013e3181a347ab. PMID 19440130
- [Background] Harris SR. A study of a dynamic proximal stability splint in the management of children with cerebral palsy. Dev Med Child Neurol. 1996 Feb;38(2):181-3. No abstract available. PMID 8603786
- [Background] Blair E, Ballantyne J, Horsman S, Chauvel P. A study of a dynamic proximal stability splint in the management of children with cerebral palsy. Dev Med Child Neurol. 1995 Jun;37(6):544-54. doi: 10.1111/j.1469-8749.1995.tb12041.x. PMID 7789663
- [Background] Romeo DM, Specchia A, Sini F, Bompard S, Di Polito A, Del Vecchio A, Ferrara P, Bernabei R, Mercuri E. Effects of Lycra suits in children with cerebral palsy. Eur J Paediatr Neurol. 2018 Sep;22(5):831-836. doi: 10.1016/j.ejpn.2018.04.014. Epub 2018 May 3. PMID 29802022
- [Background] Belizon-Bravo N, Romero-Galisteo RP, Cano-Bravo F, Gonzalez-Medina G, Pinero-Pinto E, Luque-Moreno C. Effects of Dynamic Suit Orthoses on the Spatio-Temporal Gait Parameters in Children with Cerebral Palsy: A Systematic Review. Children (Basel). 2021 Nov 5;8(11):1016. doi: 10.3390/children8111016. PMID 34828729
- [Background] Romeo DM, Bompard S, Cocca C, Serrao F, De Carolis MP, Zuppa AA, Ricci D, Gallini F, Maddaloni C, Romagnoli C, Mercuri E. Neonatal neurological examination during the first 6h after birth. Early Hum Dev. 2017 May;108:41-44. doi: 10.1016/j.earlhumdev.2017.03.013. Epub 2017 Apr 5. PMID 28390243
- [Background] Als H, Duffy FH, McAnulty GB, Rivkin MJ, Vajapeyam S, Mulkern RV, Warfield SK, Huppi PS, Butler SC, Conneman N, Fischer C, Eichenwald EC. Early experience alters brain function and structure. Pediatrics. 2004 Apr;113(4):846-57. doi: 10.1542/peds.113.4.846. PMID 15060237
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Background] Romeo DM, Cowan FM, Haataja L, Ricci D, Pede E, Gallini F, Cota F, Brogna C, Vento G, Romeo MG, Mercuri E. Hammersmith Infant Neurological Examination for infants born preterm: predicting outcomes other than cerebral palsy. Dev Med Child Neurol. 2021 Aug;63(8):939-946. doi: 10.1111/dmcn.14768. Epub 2020 Dec 18. PMID 33336801
- [Background] Turner-Stokes L. Goal attainment scaling (GAS) in rehabilitation: a practical guide. Clin Rehabil. 2009 Apr;23(4):362-70. doi: 10.1177/0269215508101742. Epub 2009 Jan 29. PMID 19179355
- [Background] Brown G. NICU noise and the preterm infant. Neonatal Netw. 2009 May-Jun;28(3):165-73. doi: 10.1891/0730-0832.28.3.165. PMID 19451078
- [Background] Lester BM, Andreozzi-Fontaine L, Tronick E, Bigsby R. Assessment and evaluation of the high risk neonate: the NICU Network Neurobehavioral Scale. J Vis Exp. 2014 Aug 25;(90):3368. doi: 10.3791/3368. PMID 25177897
- [Background] Einspieler C, Prechtl HF. Prechtl's assessment of general movements: a diagnostic tool for the functional assessment of the young nervous system. Ment Retard Dev Disabil Res Rev. 2005;11(1):61-7. doi: 10.1002/mrdd.20051. PMID 15856440